CLINICAL TRIAL: NCT03495284
Title: The Effect of Potatoes on Markers of Cardiometabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PKE POTATO
Record Dates: First submitted 2018-01-15; First posted 2018-04-11 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potato treatment (Experimental): Participants will be provided with one potato-based side dish, equivalent to one medium sized potato, every day for 4 weeks for incorporation into their self-selected diet. The potato-based side dish will be prepared at the Penn State Metabolic Kitchen. The potato side dish will consist of commonly consumed potato-based sides in the U.S. and there will be limited inclusion of ingredients high in saturated fat, refined sugars or sodium. French fries will not be provided. The variety of potatoes will represent consumption patterns in the U.S. including white, russet, yellow and red potatoes.
  Interventions: Dietary Supplement: Potato-based side dish
- Refined grain treatment (Active Comparator): Participants will be provided with a calorie-matched refined grain-based side dish every day for 4 weeks for incorporation into their self-selected diet. The refined grain-based side dishes will be prepared at the Penn State Metabolic Kitchen and ingredients high in saturated fat, refined sugar or sodium will not be used. These will be sides commonly eaten in the U.S. (e.g. pasta made with white flour and white rice, white bread rolls). During this treatment, participants will be told not to consume potatoes.
  Interventions: Dietary Supplement: Refined grain-based

INTERVENTIONS:
Dietary Supplement: Potato-based side dish — Daily consumption of a potato-based side dish equivalent to one medium size potato for 4 weeks
  Arms: Potato treatment
Dietary Supplement: Refined grain-based — Daily consumption of an isocaloric refined grain-based side dish for 4 weeks
  Arms: Refined grain treatment

SUMMARY:
A 2-period randomized cross-over trial will be conducted to determine the effect of incorporating 1 medium size potato, compared to an isocaloric portion of refined grains, on fasting glucose levels, insulin sensitivity, blood pressure, lipids and lipoproteins, arterial stiffness, body weight, gut microbiome, and dietary intake.

DETAILED DESCRIPTION:
A 2-period randomized cross-over study will be conducted. Free-living subjects will be provided with a potato based side dish (equivalent to one medium sized potato) or an isocaloric refined grain based side dish every day for 4 weeks, in random order. The treatment periods will be separated by a minimum two-week break. Endpoint testing will be conducted over two days at baseline and the end of each diet period.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* BMI > 20 and <40 kg/m2
* Male or female

Exclusion Criteria:

* Diagnosed diabetes or fasting glucose >126 mg/dl
* Hypertension (systolic blood pressure >160mmHg or diastolic blood pressure >100mmHg)
* Prescribed anti-hypertensive, lipid lowering or glucose lowering drugs
* Established cardiovascular disease, stroke, diabetes, liver, kidney or autoimmune disease or inflammatory conditions
* Use of supplements (psyllium, fish oil, soy lecithin, phytoestrogens) and botanicals and not willing to cease for the duration of the study
* Pregnancy or lactation
* Weight loss of >=10% of body weight within the 6 months prior to enrolling in the study
* Smoking or use of any tobacco products

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2020-01-19 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose | 4 weeks

SECONDARY OUTCOMES:
Homeostasis Model of Assessment of Insulin Resistance | 4 weeks
Peripheral blood pressure | 4 weeks
Central blood pressure | 4 weeks
Total cholesterol | 4 weeks
Pulse Wave Velocity | 4 weeks
Augmentation index | 4 weeks
Diet quality measured by the Healthy Eating Index 2010 | 4 weeks
Change in fecal short chain fatty acid levels | Week 0; Week 2 of treatment period 1; Week 4 of treatment period 1; Week 2 of treatment 2; Week 4 of treatment 4
Change in microbiome composition | Week 0; Week 2 of treatment period 1; Week 4 of treatment period 1; Week 2 of treatment 2; Week 4 of treatment 4
LDL cholesterol | 4 weeks
HDL cholesterol | 4 weeks
Triglycerides | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No